CLINICAL TRIAL: NCT00002567
Title: PHASE II STUDY EVALUATING AUTOLOGOUS PERIPHERAL BLOOD PROGENITOR CELL TRANSPLANTATION FOR ACUTE LEUKEMIAS
Brief Title: High-Dose Chemotherapy and Radiation Therapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Acute Leukemia in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 93-161; CDR0000063595 (Registry Identifier: PDQ (Physician Data Query)); NCI-H94-0460
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Bone Marrow Ablation; Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); bone marrow ablation; adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Filgrastim; Etoposide; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: etoposide
Procedure: peripheral blood stem cell transplantation
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose radiation therapy and etoposide followed by peripheral stem cell transplantation in treating patients with acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of myeloablative total-body irradiation and etoposide followed by autologous peripheral blood stem cell (PBSC) transplantation in prolonging the disease-free survival of patients with acute leukemia. II. Investigate the ability of growth factor-primed PBSC to provide hematopoietic reconstitution following myeloablative therapy.

OUTLINE: Patients are treated on Regimen A, then Regimen B. Regimen A: Stem Cell Mobilization. Granulocyte Colony Stimulating Factor (Amgen), G-CSF, NSC-614629. Regimen B: Radiotherapy and Myeloablative Chemotherapy with Hematopoietic Rescue. Total-Body Irradiation, TBI (high-energy electrons used for lung boost); and Etoposide, VP-16, NSC-141540; with Peripheral Blood Stem Cells, PBSC; G-CSF.

PROJECTED ACCRUAL: Up to 45 patients will be studied over approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously diagnosed acute leukemia in one of the following categories: Acute myelogenous leukemia (any subtype) in first or subsequent remission Ph+ acute lymphoblastic leukemia (ALL) in first or greater remission Ph- ALL in second or subsequent remission Cellular marrow with no morphologic evidence of residual leukemia within approximately 2 weeks of cryopreservation Negative CSF cytology required of ALL patients Allogeneic marrow transplant considered for patients under age 55 with a healthy HLA-identical family member available

PATIENT CHARACTERISTICS: Age: Over 16 to 65 Performance status: Not specified Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dl Renal: Creatinine no greater than 1.5 mg/dl OR Creatinine clearance at least 60 ml/min Cardiovascular: LVEF at least 50% by MUGA or normal on echocardiogram Pulmonary: DLCO at least 50% of predicted Other: HIV seronegative No uncontrolled infection Negative pregnancy test required of fertile women

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1994-03; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Maslak, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States